CLINICAL TRIAL: NCT06617026
Title: Short-Term Outcome of Medical Vs. Surgical Management Of Chronic Anal Fissure (A Randomized Controlled Trial)
Brief Title: Short-Term Outcome of Medical Vs. Surgical Management Of Chronic Anal Fissure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Waleed Ghareeb, Senior consultant and lecturer of General surgery, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #5787
Record Dates: First submitted 2024-09-20; First posted 2024-09-27 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Anal Fissure Chronic
Keywords: Chronic anal fissure
MeSH Terms: interventions — Sucralfate; azadirachtin; hyperforin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sucralfate Group (Experimental): patients assigned to this group will start to use a topical rectal ointment containing Sucralfate. The patients are instructed to apply it twice a day, using a gloved finger, inside the anal canal and the perianal region for 40 days. the follow-up visits are arranged at 15, 30 and 40 days.
  Interventions: Drug: Sucralfate
- HyperOil Group (Experimental): patients assigned to this group will start to use topical oil containing the combination of azadirachtin and hyperforin. The patients are instructed to apply it twice a day, using a gloved finger, inside the anal canal and the perianal region for 40 days. the follow-up visits are arranged at 15, 30 and 40 days.
  Interventions: Drug: Azadirachtin
- Surgery (Active Comparator): patients assigned to this group will be operated for fissurectomy and lateral sphincterectomy. the follow-up visits are arranged at 15, 30 and 40 days.
  Interventions: Procedure: fissurectomy and lateral sphincterectomy

INTERVENTIONS:
Drug: Sucralfate — a topical rectal ointment. The patients are instructed to apply it twice a day, using a gloved finger, inside the anal canal and the perianal region for 40 days
  Arms: Sucralfate Group
Drug: Azadirachtin — a topical oil. The patients are instructed to apply it twice a day, using a gloved finger, inside the anal canal and the perianal region for 40 days
  Other Names: azadirachtin and Hyperforin
  Arms: HyperOil Group
Procedure: fissurectomy and lateral sphincterectomy — fissurectomy and lateral sphincterectomy
  Arms: Surgery

SUMMARY:
Several topical agents have been proposed for Chronic anal fissure (CAF) treatment with the common goal of increasing anodermal blood flow to promote healing but approaching the use of medical treatment in CAFs is not standardized yet. Thus, the present study aimed to compare the efficacy and safety of Sucralfate (Emoflon®), the combination of azadirachtin and hyperforin (HyperOil®) and the traditional surgical treatment (lateral sphincterotomy) in patients with CAFs.

DETAILED DESCRIPTION:
Several topical agents have been proposed for Chronic anal fissure (CAF) treatment with the common goal of increasing anodermal blood flow to promote healing but approaching the use of medical treatment in CAFs is not standardized yet. Thus, the present study aimed to compare the efficacy and safety of Sucralfate (Emoflon®), the combination of azadirachtin and hyperforin (HyperOil®) and the traditional surgical treatment (lateral sphincterotomy) in patients with CAFs.

Study Objective:

Primary Objectives:

1. To evaluate the efficacy and safety of Sucralfate (Emoflon®), the combination of azadirachtin and hyperforin (HyperOil®) and the traditional surgical treatment (lateral sphincterotomy) in patients with CAFs.

Study Design:

A prospective randomized controlled trial

Study sampling:

A convenience sampling method will be used; all patients seeking medical advice for CAF at Suez Canal University hospitals, the Faculty of Medicine during the study period and fulfill the inclusion criteria will be recruited. One of the researchers who will make random allocation cards using an Excel formula algorithm will perform simple randomisation.

Methodology:

This study will include at least 99 patients with CAFs of both genders who will visit the general surgery clinic in the faculty of medicine at Suez Canal University hospital and fulfil the inclusion and exclusion starting from September 2024. Patients of both genders with CAF for the first time, above 18 years old and ASA I/II will be included in the study. While patients with sepsis, previous pelvic radiation, recurrent CAF, with malignancy, on immunosuppressive drugs, with pregnancy or lactation will be excluded. Patients will be randomly allocated into 3 groups at a ratio of 1:1:1 starting with the Sucralfate group. Formal written consent will be obtained from the study participants prior to being involved in the study. All included patients will be followed up to 40 days.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years old.
* CAFs for the first time
* ASA I, II

Exclusion Criteria:

* Sepsis
* Previous pelvic radiation.
* recurrent chronic anal fissure
* Pregnancy or lactation.
* Immunosuppressive state
* Malignancy
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
REALISE score | in each 3 follow up visits (visit 1,2, and 3 after 15, 30 , and 40 days respectively)
  REALISE (scoRing systEm for AnaL fIsSurE), will be used to assess pain (score range 0-10), quality of life, duration of pain, intake of analgesics and bleeding. The latter four items were rated on a scale of 1-5

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt